CLINICAL TRIAL: NCT04037644
Title: Effect of Volume EXpansion witH ALbumin vs. Crystalloid on EIT-derived Expiratory Lung Impedance in Critically Ill, Hemodynamically Unstable Patients. A Single-blind, Randomized and Controlled Study
Brief Title: Volume Expansion With Albumin vs. Crystalloid and Expiratory Lung Impedance
Acronym: EXHALE
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Davide Chiumello, Director of Intensive Care, University of Milan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EXHALE
Record Dates: First submitted 2019-07-24; First posted 2019-07-30 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Circulatory Failure
MeSH Terms: conditions — Shock | interventions — Albumins; Ringer's Lactate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Albumin (Experimental): fluid loading with 200 mL of 4% albumin over a 10' interval
  Interventions: Procedure: Fluid loading with Albumin
- Ringer Lactate (Active Comparator): fluid loading with 5 mL/kg actual body weight of Ringer Lactate over a 10' interval
  Interventions: Procedure: Fluid loading with Ringer Lactate

INTERVENTIONS:
Procedure: Fluid loading with Albumin — Fluid loading with 200 ml of 4% Albumin to reverse acute circulatory failure
  Arms: Albumin
Procedure: Fluid loading with Ringer Lactate — Fluid loading with 5 ml per kg of actual body weight to reverse acute circulatory failure
  Arms: Ringer Lactate

SUMMARY:
Acute circulatory failure reduces oxygen delivery below cellular requirements, potentially leading to organ failure. Intravenous fluids are generally administered with the aim of increasing cardiac output and restore organ perfusion. Nevertheless, only 50% of patients increase their cardiac output, while in the remainder not only does fluid loading provide no benefit but it also leads to volume overload (peripheral and pulmonary edema).

There are two types of resuscitation fluids, colloids and crystalloids. Given their oncotic pressure, colloids should remain in the intravascular space, while crystalloids distribute into the whole extracellular compartment, potentially increasing the risk of tissue edema. Surprisingly, only few studies directly compared albumin and crystalloids in terms of their overload-related side effects.

Electrical impedance tomography (EIT) is a noninvasive, radiation-free, lung imaging modality, which shows lung impedance as determined by small electrical currents. An increase in intrapulmonary gas volume increases impedance, while an increase in blood or fluid volume, lowers it. EIT has a high temporal resolution, allowing to assess ventilation and perfusion in real-time. Preliminary data suggest its value to assess the variations of intrathoracic fluid in patients with pulmonary edema.

The aim of the present single-blind, randomized, controlled study is to compare the effect of a fluid challenge with albumin vs. crystalloids on EIT-derived lung impedance in a group of 56 critically ill patients with acute circulatory failure. Our hypothesis is that fluid challenge with albumin leads to a lesser decrease in lung impedance, that is a lesser extravasation of fluids into the lungs.

Hemodynamic and respiratory variables, blood samples, cardiac ultrasound and EIT measurements will be recorded before the fluid challenge, and repeated at the end of fluid infusion, 20 and 60 minutes after. Factorial Analysis of variance for repeated measures will be used to assess the effects of fluid loading

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years with acute circulatory failure of any cause, receiving mechanical ventilation using volume-assisted control mode, without any spontaneous breathing activity, scheduled for a fluid bolus by their treating physician will be enrolled. Patients will only be included in the study once.

Acute circulatory failure will be defined as the presence of a systolic blood pressure (SBP) ≤90 mmHg or mean arterial pressure (MAP) ≤70 mmHg or requiring vasopressors to maintain SBP >90 mmHg or MAP >70 mmHg, along with one or more of the following: 1) urinary flow ≤0.5 mL/kg/h for ≥2 hours, 2) heart rate ≥100 beats per minute, 3) presence of skin mottling, 4) blood lactate concentration ≥2 mmol/L, 5) oxygen saturation in the central venous blood <65%.

Exclusion Criteria:

* Patients having right ventricular dysfunction, anuria, pregnancy, presence of pneumothorax or lung emphysema, previous history of severe chronic obstructive pulmonary disease (GOLD III-IV) or contraindications to the use of EIT (e.g., presence of pacemaker or automatic implantable cardioverter-defibrillator) and impossibility to place the EIT belt in the right position (e.g., presence of surgical wounds dressing) will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2019-07-24 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in lung impedance | Day 1
  Reduction in EIT-derived end-expiratory lung impedance after the fluid challenge in the group of patients who will receive albumin as compared to patients who will receive crystalloids

SECONDARY OUTCOMES:
Comparison of the change expiratory lung impedance, as assessed by EIT, in fluid responders and non-responders | Day 1
  Comparison of the change in end-expiratory lung impedance, as assessed by EIT, after the fluid challenge with albumin or Ringer Lactate, in patient who will respond to the fluid challenge with an increase in their stroke volume, as compared to those who will not (non-responders)
Effect of fluid loading with albumin or Ringer Lactate on the change in arterial blood oxygenation | Day 1
  Assesment of the reduction in oxygenation, as assessed by blood gas analysis, after the fluid challenge in the group of patients who will receive albumin as compared to patients who will receive crystalloids, and its relationship with the change in expiratory lung impedance, as assessed by EIT

CONTACTS AND LOCATIONS:
Overall Officials: Davide Chiumello, MD, Principal Investigator — Ospedale San Paolo - Polo Universitario, ASST Santi Paolo e Carlo, Milan
Locations (1):
- Ospedale San Paolo - Polo Universitario, ASST Santi Paolo e Carlo, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: No